CLINICAL TRIAL: NCT03388840
Title: the Effect of Adipose Derived Stem Cells Combined With Platelet Rich Plasma Versus Platelet Rich Plasma Alone on Follicular Unit Extraction Hair Transplantion in Male Androgenic Alopecia: Clinical Trial
Brief Title: Adipose Derived Stem Cells Versus Platelet Rich Plasma on Follicular Unit Extraction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, A Ghazally, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADSCPRPFUE
Record Dates: First submitted 2017-12-23; First posted 2018-01-03 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-02

CONDITIONS: Androgenetic Alopecia
Keywords: platelet rich plasma; adipose derived stem cells; follicular unit extraction; hair transplantation
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adipose derived stem cells suspention (Experimental): suspension rich in adipose derived stem cells plus platelet rich plasma will be injected at the recipient site during follicular unit extraction for treatment of androgenetic alopecia
  Interventions: Biological: Adipose derived stem cells suspention
- Platelet rich plasma (Active Comparator): platelet rich plasma will be injected at the recipient site during follicular unit extraction for treatment of androgenetic alopecia
  Interventions: Biological: Platelet rich plasma

INTERVENTIONS:
Biological: Adipose derived stem cells suspention — application of adipose derived stem cells to the engrafted hair in hair transplantation surgery
  Arms: Adipose derived stem cells suspention
Biological: Platelet rich plasma — application of autologous platelet rich plasma to the engrafted hair in hair transplantation surgery
  Arms: Platelet rich plasma

SUMMARY:
Androgenetic alopecia is the most common type of alopecia in both men and women. About 80 % of Caucasian men and 40-50 % of Caucasian women are affected by androgenetic alopecia. The psychological impact of hair loss due to Androgenetic alopecia can be profound.

DETAILED DESCRIPTION:
Currently, two medications are Food and Drug Administration approved in the treatment of Androgenetic alopecia which are minoxidil, and finasteride. Both medications must be taken indefinitely for benefits to persist. Hair transplantation is the only current successful permanent option. Nowadays, the majority of surgeons use 2 techniques, the classic strip technique, and the follicular unit extraction technique. Advantages of follicular unit extraction over the strip technique are the lesser incidence of donor zone post-procedural discomfort and the barely visible scarring.

Platelet rich plasma is an autologous concentration of platelets in small volume of plasma and is an exciting therapeutic option for hair growth. Combining platelet rich plasma with follicular unit extraction surgery for the treatment of Androgenetic alopecia demonstrated that PRP is able to minimize the postsurgical follicle loss and potentiate the performance of grafted hairs.

Adipose derived stem cells are an effective mesenchymal stem cell population with enormous potential in different fields of regenerative medicine.

Adipose stem cells are needed to induce the proliferation of bulge stem cells of hair follicle. Furthermore, they can help in wound healing and vascular neogenesis.

Zanzottera et al. 2014 investigated the effect of adipose derived stem cells on wound healing and engraftment of the transplanted hair applied during hair restoration surgery for three patients with androgenetic alopecia. Despite their promising results, further clinical trials including larger number of patients are still needed to confirm their preliminary findings.

ELIGIBILITY:
Inclusion Criteria:

* male patients with androgenetic alopecia between 18 years and 60 years

Exclusion Criteria:

1. Patients with Non-androgenetic causes of hair loss.
2. Female patients with androgenetic alopecia.
3. Patients who received anti-hair loss treatment within the past six months.
4. Patients with history of bleeding disorders or on anticoagulant therapy.
5. Patients with history of chronic liver disease, cancer or connective tissue disorders.
6. Patients with current scalp infection.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
hair growth | 12 months
  Evaluate the effect of adipose derived stem cells intradermally injected in the recipient site during follicular unit extraction for the treatment of androgenetic alopecia on transplanted hair growth in terms of hair density (number of hairs / cm2) in the transplanted region using folliscope.

SECONDARY OUTCOMES:
hair shaft diameter | 12 months
  Evaluate the effect of adipose derived stem cells intradermally injected in the recipient site during follicular unit extraction for the treatment of androgenetic alopecia on transplanted hair shaft diameter in mm using folliscope.

CONTACTS AND LOCATIONS:
Overall Officials: Alaa H Ghazally, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospitals, Asyut, Egypt

REFERENCES:
- [Background] Adil A, Godwin M. The effectiveness of treatments for androgenetic alopecia: A systematic review and meta-analysis. J Am Acad Dermatol. 2017 Jul;77(1):136-141.e5. doi: 10.1016/j.jaad.2017.02.054. Epub 2017 Apr 7. PMID 28396101
- [Background] Navarro RM, Pino A, Martinez-Andres A, Molina C, Martinez AM, Martinez N, Orive G, Anitua E. The effect of plasma rich in growth factors combined with follicular unit extraction surgery for the treatment of hair loss: A pilot study. J Cosmet Dermatol. 2018 Oct;17(5):862-873. doi: 10.1111/jocd.12446. Epub 2017 Oct 26. PMID 29076290
- [Background] Jimenez-Acosta F, Ponce-Rodriguez I. Follicular Unit Extraction for Hair Transplantation: An Update. Actas Dermosifiliogr. 2017 Jul-Aug;108(6):532-537. doi: 10.1016/j.ad.2017.02.015. Epub 2017 May 5. English, Spanish. PMID 28483047
- [Background] Qi J, Garza LA. An overview of alopecias. Cold Spring Harb Perspect Med. 2014 Mar 1;4(3):a013615. doi: 10.1101/cshperspect.a013615. PMID 24591533